CLINICAL TRIAL: NCT02850029
Title: An International Survey on Aminoglycoside Practices in Critically Ill Patients: AMINO III Survey
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: IRB 15 04 08
Record Dates: First submitted 2016-07-27; First posted 2016-07-29 (Estimated); Last update posted 2025-11-21 (Actual); Status verified 2019-01

CONDITIONS: Underdosing of Aminoglycosides; Critical Illness
Keywords: antimicrobial; intensive care units
MeSH Terms: conditions — Critical Illness | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- critically ill patients: Critically ill patients admitted in intensive care units and receiving one of the following aminoglycosides: gentamicin, tobramycin and amikacin as part of their usual care.
  Interventions: Other: Observational study, no intervention

INTERVENTIONS:
Other: Observational study, no intervention

SUMMARY:
This is an international observational cohort study on current aminoglycoside practices in intensive care units. Clinical and demographic data, dosing and therapeutic drug monitoring data will be collected during the first week of aminoglycoside (tobramycin, amikacin or gentamicin) administration in different countries over a year. A minimum of ten consecutive patients will be enrolled at each site.

DETAILED DESCRIPTION:
Aminoglycosides are commonly used antibiotics for difficult to treat infections. However, aminoglycoside administration varies widely among countries. The aim of this multicenter observational study is to provide up-to-date and comprehensive descriptive data on current aminoglycoside (tobramycin, amikacin or gentamicin) use in a large cohort of critically ill patients in different countries. The benefits expected from this study are a better understanding of worldwide aminoglycoside prescription variability in critically ill patients and to determine the risk factors of inadequate aminoglycoside dosing regimens.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Intensive care unit patients
* Receiving aminoglycoside therapy for a sepsis according to the Third International Consensus Definitions for Sepsis and Septic Shock

Exclusion Criteria:

* Aged < 18 years of age
* Previous inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Large cohort of intensive care units patients receiving aminoglycosides (tobramycin, amikacin or gentamicin) as part of their antimicrobial therapy for sepsis.
Sampling Method: Non-Probability Sample
Enrollment: 964 (Actual)
Dates: Start 2016-05-21 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Aminoglycoside current practices descriptive data in intensive care units | Seven first days of aminoglycoside therapy

SECONDARY OUTCOMES:
Aminoglycoside dosing regimens | Seven first days of aminoglycoside therapy
Aminoglycoside therapy duration | Seven first days of aminoglycoside therapy
Aminoglycoside therapeutic drug monitoring | Seven first days of aminoglycoside therapy

CONTACTS AND LOCATIONS:
Overall Officials: Claire Roger, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (84):
- Australia (5):
  - Royal Brisbane Women's Hospital, Brisbane, Queensland
  - Royal Brisbane and Women's Hospital, Brisbane
  - Frankston Hospital Victoria, Frankston
  - Sunshine Coast hospital, Sunshine Coast
  - Toowoomba Hospital, Toowoomba
- Chile (4):
  - Hospital Base de Valvidia, Valdivia, Los Ríos Region
  - Hospital Barros Luco Trudeau, Santiago
  - Hospital CU Chile, Santiago
  - Salvador Santiago Hospital, Santiago
- France (61):
  - APHM La timone, Marseille, PACA
  - Centre Hospitalier Aix-En-Provence, Aix-en-Provence
  - Centre Hospitalier D'Ales, Alès
  - Chu Amiens, Amiens
  - Chu Angers, Angers
  - Centre Hospitalier Arles, Arles
  - CHI Robert Ballanger, Aulnay-sous-Bois
  - Centre Hospitalier Aurillac, Aurillac
  - Centre Hospitalier Avignon, Avignon
  - Chru Besancon, Besançon
  - Chu Bordeaux, Bordeaux
  - Centre Hospitalier de BOULOGNE SUR MER, Boulogne-sur-Mer
  - Centre Hospitalier Bourg En Bresse, Bourg-en-Bresse
  - Chru Brest, Brest
  - Chu Brest- Hopital Cavale, Brest
  - CHU CAEN, Caen
  - Centre Hospitalier Charleville-Mezieres, Charleville-Mézières
  - Chu Clermont-Ferrand, Clermont-Ferrand
  - Centre Hospitalier de Compiegne, Compiègne
  - Chu Grenoble, Grenoble
  - Centre Hospitalier La Rochelle-Hopital Saint Louis, La Rochelle
  - Centre Hospitalier du Mans, Le Mans
  - Chu Lyon- Hopital La Croix Rousse, Lyon
  - Chu Lyon- Lyon Sud, Lyon
  - Aphm- La Conception, Marseille
  - AP-HM - Hopital Nord, Marseille
  - Centre Hospitalier Sambre-Avesnois, Maubeuge
  - Centre Hospitalier de Montauban, Montauban
  - CHU MONTPELLIER-Hopital Lapeyronnie, Montpellier
  - CHU MONTPELLIER-Hopital St Eloi, Montpellier
  - Centre Hospitalier de MORLAIX, Morlaix
  - Chru Nancy -Hopital de Brabois, Nancy
  - Chu Nantes- Hopital Hotel Dieu, Nantes
  - CHU NANTES- hôpital Nord Laennec, Nantes
  - CHU Nice- Hopital Pasteur, Nice
  - CHU Nice-Hopital L'Archet, Nice
  - Centre Universitaire de Nimes, Nîmes
  - AP-HP - Paris St Louis, Paris
  - AP-HP - Hopital Paris St Antoine, Paris
  - Aphp - Pitie Salpetriere, Paris
  - Aphp- Pitie Salpetriere, Paris
  - APHP- Bichat, Paris
  - APHP- Descartes, Paris
  - APHP-Hopital Georges Pompidou, Paris
  - AP-HP - Bicetre, Paris
  - Centre Hospitalier de PAU, Pau
  - Chu Poitiers, Poitiers
  - CHU REIMS- Hopital Robert Debré, Reims
  - CHU RENNES - Hopital Pontchaillou, Rennes
  - Centre Hospitalier de Roanne, Roanne
  - Centre Hospitalier de Rodez, Rodez
  - CHU ROUEN- Hopital Nicolle, Rouen
  - Centre Hospitalier Sainte Catherine, Saint-Brieuc
  - CHU La Reunion-Hopital Felix Guyon, Saint-Denis
  - CHU SAINT-ETIENNE - Hopital Nord, Saint-Etienne
  - Centre Hospitalier de Salon de Provence, Salon-de-Provence
  - Centre Hospitalier Sainte Catherine, Saverne
  - Centre Hospitalier de Toulon, Hopital Sainte Musse, Toulon
  - CHU TOULOUSE- Hopital Rangueil, Toulouse
  - Centre Hospitalier Valence, Valence
  - Centre Hospitalier de Valenciennes, Valenciennes
- Greece (5):
  - Athens Hippocratio Hospital, Athens
  - Naval and Veterans Hospital of Athens, Athens
  - University Critical Care Department Aghioi Anargyroi Hospital, Athens
  - University Hospital of loannina, Ioannina
  - G. Gennimatas General Hospital, Thessaloniki
- United Kingdom (9):
  - Sandwell and west Birmingham hospital, Birmingham
  - University Hospital Birmingham, Birmingham
  - Guy'S and St Thomas', London
  - Salford royal, Manchester
  - University Hospital of South Manchester, Manchester
  - Oxford Radcliffe Hospitals, Oxford
  - St Helens and Knowsley Hospitals, Prescot
  - Sheffield Teaching Hospitals, Sheffield
  - Southampton University Hospitals, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Roger C, Louart B, Elotmani L, Barton G, Escobar L, Koulenti D, Lipman J, Leone M, Muller L, Boutin C, Amour J, Banakh I, Cousson J, Bourenne J, Constantin JM, Albanese J, Roberts JA, Lefrant JY; Azurea Network. An international survey on aminoglycoside practices in critically ill patients: the AMINO III study. Ann Intensive Care. 2021 Mar 19;11(1):49. doi: 10.1186/s13613-021-00834-4. PMID 33740157